CLINICAL TRIAL: NCT05541770
Title: Assessment of Multidisciplinary Clinics Implementation in Cancer Patients' Management in Arab Countries
Brief Title: Application of MDT Clinics in Arab World
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Riham H. AbdelAziz, Clinical Oncology Lecturer and consultant, Cairo University
Other Study IDs: Oncosurvey
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Multidisciplinary Communication
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Healthcare workers/Physicians involved in cancer diagnosis & management in the Arab countries should respond to a survey

SUMMARY:
Multidisciplinary clinics affect the quality of management of cancer patients. This Questionnaire is for research purposes aiming at exploring the application and implementation of multidisciplinary clinics in managing cancer patients in the Arab countries. The results of this survey will shed the light on the situation; the investigators aim at exploring the status of their implementation and who participates in them, in addition to exploring the challenges that face MDT clinics in Arab world.

DETAILED DESCRIPTION:
Multidisciplinary teams (MDTs) are recommended as a corner stone of best cancer care nowadays. MDTs consist of many professionals such as medical, nursing, and allied professionals and diagnostic experts to determine the optimal treatment pathway for individual patients. They should be well organized and efficient. MDT clinics care is helpful in making clinical decision and improving the quality of patients' care. However, there are many challenges that face the actual implementation and application of MDT clinics in routine cancer patients' care in our Arab countries.

This study aims at describing the situation in our Arab countries and reflecting the pathway & logistics of referring cancer patients to MDT & the impact of that on the patients' management & outcome, in addition to exploring the challenges that face effective implementation of MDT clinics, so that it can lead the improvement in oncology manangement

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers/Physicians involved in cancer diagnosis & management in the Arab countries.

Exclusion Criteria:

* Health care workers/ Physicians who are not entitled for cancer management.
* Physicians who are not working in the Arab counties.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Oncology or non oncology physicians across the Arab countries.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Investigate the rate of discussing the suspected patients in MDT clinics | Two months
  We would like to know the rate of discussing suspected patients in MDT clinics. This will be done via a questionnaire.
Investigate the main challenges to establish effective MDT clinics. | Two months
  We would like to know the main challenges to establish effective MDT clinics according to the physicians' point of view, who attend the MDT clinics . This will be done via a questionnaire.

SECONDARY OUTCOMES:
Describe the rate of well established and effective MDT in the Arab countries. | Two months
  We would like to know the rate of the well established MDT clinics and discussion during cancer patients' management. This will be done via a questionnaire.
Who usually attend the MDT in the Arab countries? | Two months
  We would like to know who usually participate and attend the MDT clinics during cancer patients' management. This will be done via a questionnaire.

IPD SHARING:
Plan to Share IPD: Undecided
This Questionnaire is for research purposes aiming at exploring the application of multidisciplinary clinics in managing our cancer patients in the Arab countries and highlighting the challenges faced by oncologists trying to establish effective MDT clinics.The data will be published when completed.